CLINICAL TRIAL: NCT03098316
Title: Metabolomics in Surgical Ophthalmological Patients
Acronym: MISO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: FRO (Funds for Research in Ophthalmology, Belgium) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Stalmans Ingeborg, Head of the glaucoma department, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: MISO Study
Record Dates: First submitted 2017-03-26; First posted 2017-03-31 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Primary Open-angle Glaucoma; Low Tension Glaucoma
Keywords: Cross sectional studies; Metabolomics; Glaucoma; Low tension glaucoma; Ophthalmologic surgical procedures
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma, urine, aqueous humor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- POAG: Primary open angle glaucoma patients
  Interventions: Diagnostic Test: Metabolomics analysis of patient samples
- NTG: Normal/Low tension glaucoma patients
  Interventions: Diagnostic Test: Metabolomics analysis of patient samples
- Control: Patients with cataract and without glaucoma or other eye diseases
  Interventions: Diagnostic Test: Metabolomics analysis of patient samples

INTERVENTIONS:
Diagnostic Test: Metabolomics analysis of patient samples — Metabolomics analysis of patient samples by mass spectrometry and nuclear magnetic resonance spectroscopy.

SUMMARY:
Metabolomics consists in the study of metabolites in body fluids or tissues. It investigates the consequences of the activity of genes and proteins. One of its advantages is that it is able to do a simultaneous measurement of metabolic changes in living organisms as a response to a disturbance (disease, diet, environment, others) and because a metabolic profile is summative of all the biochemical processes occurring in the body at a given time, it makes no presumption about the relative importance of these processes. Ultimately it is a fingerprint of the organism's health status, at a given time.

Metabolomic analysis of serum, plasma and urine has revealed panels of metabolites that distinguish patients with cardiovascular disease, breast cancer, Parkinson disease, Alzheimer's disease and diabetes from control patients. Regarding ocular diseases only few studies have been published, related to diabetic retinopathy, retinal detachment, age-related macular degeneration, uveitis and glaucoma.

Glaucoma is one of the leading causes of blindness in the world, according to the World Health Organization, and there are still no biomarkers that can provide an early diagnosis. Nowadays, glaucoma classification relies substantially in the measurement of intraocular pressure (IOP), which can be rather artificial and also unreliable since IOP values can fluctuate during the day. Moreover, patients with normal IOP values can also develop glaucomatous neuropathy (normal-tension glaucoma, NTG) and progress even when IOP is decreased. Several studies have shown that NTG patients suffer from a systemic vascular dysregulation, with higher rates of systemic hypotension, Raynaud phenomenon and migraine. Hence, other mechanisms than an increased IOP are of importance in the development and progression of glaucoma.

Only one metabolome-wide study has been made in glaucoma (Burgess, I.; 2015). In a sample of 72 american patients with primary open angle glaucoma (POAG), the authors found significant differences in comparison to controls.

The hypothesis for this study is that glaucoma patients will differ from controls, and POAG patients will differ from NTG patients. The investigators will look into metabolomics as a way to create a method to diagnose and stratify patients, as an add-on or alternative to the currently available diagnostic tools like IOP, functional and structural measurement.

DETAILED DESCRIPTION:
This is a cross sectional study built to compare samples from glaucoma patients undergoing surgery (open-angle glaucoma and normal-tension glaucoma, age and gender matched) with age and gender-matched controls (healthy patients undergoing cataract surgery). For this the investigators will collect plasma, urine and aqueous humor to be analyzed through mass spectrometry and nuclear magnetic resonance spectroscopy. Patients have a night fasting period prior to sample collection, and a lifestyle and food frequency questionnaire is filled to control for nutritional influence on metabolites. Diabetic patients are excluded, since it would confound our analysis.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patients (POAG/NTG): undergoing trabeculectomy, XEN® implantation or cataract surgery
* Controls (non glaucoma): undergoing cataract surgery
* Caucasian

Exclusion Criteria:

* Diabetes mellitus
* any intra ocular surgery on study eye, other than clear cornea cataract surgery more than one year before
* other eye pathologies than the one the surgery is intended for (except refractive error and cataract in glaucoma patients), namely retinopathies, uveitis and other causes for neuropathy.

Ages: 60 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients from the ophthalmology department that are undergoing intraocular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Metabolomics profile of each group | Morning of the surgery
  un-targeted metabolomics and identification of metabolites based on exact mass using metabolomics library

SECONDARY OUTCOMES:
Surgical success of glaucoma patients | 12 months
  Success is defined as an IOP between 6 and 18 mmHg with a reduction of 30% from baseline, and was sub-categorized as complete success if accomplished without glaucoma medication, qualified success with glaucoma medication, and total success as a combination of both complete and qualified. Eyes needing further glaucoma surgery, IOP ≤5 or > 18 mmHg on two consecutive visits, or loss of light perception due to glaucoma were considered as failures. Needling of encysted blebs is not considered a failure.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided